CLINICAL TRIAL: NCT01106274
Title: Study of the Effects of Riboflavin/ Ultraviolet-A Corneal Cross-linking
Brief Title: The Effects of Riboflavin/ Ultraviolet-A Corneal Cross-linking on the Signs and Symptoms of Bullous Keratopathy
Acronym: C3R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUMS-88191
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2008-10

CONDITIONS: Bullous Keratopathy
MeSH Terms: interventions — PUVA Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: ultraviolet-A — Corneal cross linking (C3R) with riboflavin and ultraviolet-A (UVA, 370 nm, 3mW/cm2) for 30 min

SUMMARY:
Recently, riboflavin (0.1%) and ultraviolet-A (UVA) collagen cross-linking (C3R) has shown potential to improve the signs and symptoms of bullous keratopathy .The objective of this study is to demonstrate the effects of C3R to treat bullous keratopathy.

ELIGIBILITY:
Inclusion Criteria:

* patients with bollous keratopathy

Exclusion Criteria:

* corneal scarring or contemporary eye disease affecting VA were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Study Completion 2009-09 (Actual)